CLINICAL TRIAL: NCT03350581
Title: Does the Merged 3D Imaging Improve Contact Force and Long Term Procedure Outcome in Atrial Fibrillation? (MICRO-AF Study)
Brief Title: Does the Merged 3D Imaging Improve Contact Force and Long Term Procedure Outcome in Atrial Fibrillation?
Acronym: MICRO-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Hong Euy Lim, MD, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUGH17237 (MICRO-AF)
Record Dates: First submitted 2017-11-15; First posted 2017-11-22 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation; Fast anatomical mapping (FAM); Computed tomography (CT); Magnetic resonance image (MRI); Contact force; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAM-CT 3D map group (Active Comparator): Operator will perform radiofrequency catheter ablation using 3D map which is constructed by integration of FAM with CT or MRI.
  Interventions: Procedure: FAM-CT 3D map group
- FAM 3D map group (Experimental): Operator will perform radiofrequency catheter ablation using 3D map which is constructed by integration of FAM alone.
  Interventions: Procedure: FAM 3D map group

INTERVENTIONS:
Procedure: FAM 3D map group — Radiofrequency catheter ablation using the 3D map which is constructed by FAM alone.
  Arms: FAM 3D map group
Procedure: FAM-CT 3D map group — Radiofrequency catheter ablation using the 3D map which is constructed by the integration of the FAM with CT or MRI.
  Arms: FAM-CT 3D map group

SUMMARY:
The purpose of the study is to investigate whether or not there are the differences in acute procedure and long-term clinical outcome of radiofrequency catheter ablation (RFCA) for atrial fibrillation (AF) using the 3D map constructed by the integration of CT(or MRI) with the fast anatomical mapping (FAM) versus using the 3D map constructed by FAM only.

DETAILED DESCRIPTION:
In a recent study, ablation therapy of AF was superior to antiarrhythmic drug therapy alone in preventing atrial arrhythmia recurrences in patients with paroxysmal or persistent AF. Various techniques have been proposed and are currently under investigation in various electrophysiology laboratories, with increasing knowledge of the pathophysiology of human AF and critical assessment of clinical outcome after the procedure. The factors related with the technical success involves appropriate contact force between catheter tip and target tissue for the complete electrical blockade and transmural ablation scar formation through continuous and sufficient energy transfer.

For improving contact and energy transfer, it is required to accurately visualize the 3D anatomy of the left atrium in order to reduce fluoroscopic exposure during the procedure. For the purpose, electro-anatomic mapping systems (EAM) are commonly being used to reconstruct a virtual 3D chamber anatomy through the acquisition of a limited number of anatomical surface location points derived from the position of the catheter tip and an extrapolation of the chamber surface in between these acquired anatomical points.

Previously, a more detailed appreciation of the complex left atrium (LA) anatomy can be obtained with 3D-anatomical chamber reconstructions derived from the computed tomography (CT) or magnetic resonance imaging(MRI). Integration of EAM with CT (or MRI) was generally regarded as a more accurate method. However, the method needs to be improved since it sometimes generates significant error during the integration process. Recently, volume-rendered 3D imaging can be created more accurately and easily through fast anatomical mapping (FAM) using multi-polar catheter. Furthermore, 3D anatomy obtained by FAM might provide more sophisticated information than that obtained from CT or MRI images since it reflects the real-time physiology and shape of the heart during the ablation procedure.

However, there have been no prospective studies investigating that 3D anatomy obtained through which method can help to improve acute or long-term procedural outcome of the ablation procedure as well as reduce procedure-related adverse effects or complications.

The purpose of the study is to investigate the differences between the 3D map constructed by the integration of the FAM with CT or MRI (FAM-CT 3D map) and that by FAM (FAM 3D map) alone with respect to following aspects:

1. the contact force between the electrode and the atrial tissue during the ablation procedure;
2. the safety and the procedure-related complications during or after the ablation procedure;
3. the long term procedural outcome after the ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first-time catheter ablation for AF.
* Willing and able to provide informed consent
* Age greater than or equal to 18 years.

Exclusion Criteria:

* Patients who have previously undergone AF ablation
* Patients with more than mild mitral valve stenosis or mechanical mitral valve replacement
* Patients with chronic renal impairment with creatinine clearance rate of < 50

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Freedom rate of any atrial tachy-arrhythmia at 1 year after ablation procedure | Within 1 year after the ablation procedure
  Any recurrence of ECG or Holter documented sustained AF >30 s duration.

SECONDARY OUTCOMES:
Contact Force distribution during procedure (g/cm2) | during procedure
  Measurements from the SmartTouch™ catheter(Biosense Webster Inc.) integrated with the Carto3®(Biosense Webster Inc.)
Rate of bidirectional conduction block | during procedur
  in linear ablation line
Percentage of pulmonary vein isolation | during procedure
  with one encircling line
Total procedural time | during procedure
  Time duration from the transseptal puncture to the end of the procedure
Total cumulative amount of radiation exposure | during procedure
  related with the procedure
Procedure-related complication rate | Within 1 year after the ablation procedure
  any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hong Euy Lim, MD, PhD, Principal Investigator — Professor
Locations (2):
- South Korea (2):
  - Korea University Guro Hospital, Seoul, Guro-gu
  - Bucheon Sejong Hospital, Bucheon-si

REFERENCES:
- [Background] Miyazaki S, Kuwahara T, Takahashi A, Kobori A, Takahashi Y, Nozato T, Hikita H, Sato A, Aonuma K, Hirao K, Isobe M. Effect of left atrial ablation on the quality of life in patients with atrial fibrillation. Circ J. 2008 Apr;72(4):582-7. doi: 10.1253/circj.72.582. PMID 18362429
- [Background] Stabile G, Bertaglia E, Senatore G, De Simone A, Zoppo F, Donnici G, Turco P, Pascotto P, Fazzari M, Vitale DF. Catheter ablation treatment in patients with drug-refractory atrial fibrillation: a prospective, multi-centre, randomized, controlled study (Catheter Ablation For The Cure Of Atrial Fibrillation Study). Eur Heart J. 2006 Jan;27(2):216-21. doi: 10.1093/eurheartj/ehi583. Epub 2005 Oct 7. PMID 16214831
- [Background] Reddy VY, Shah D, Kautzner J, Schmidt B, Saoudi N, Herrera C, Jais P, Hindricks G, Peichl P, Yulzari A, Lambert H, Neuzil P, Natale A, Kuck KH. The relationship between contact force and clinical outcome during radiofrequency catheter ablation of atrial fibrillation in the TOCCATA study. Heart Rhythm. 2012 Nov;9(11):1789-95. doi: 10.1016/j.hrthm.2012.07.016. Epub 2012 Jul 20. PMID 22820056
- [Background] Kuck KH, Reddy VY, Schmidt B, Natale A, Neuzil P, Saoudi N, Kautzner J, Herrera C, Hindricks G, Jais P, Nakagawa H, Lambert H, Shah DC. A novel radiofrequency ablation catheter using contact force sensing: Toccata study. Heart Rhythm. 2012 Jan;9(1):18-23. doi: 10.1016/j.hrthm.2011.08.021. Epub 2011 Aug 26. PMID 21872560
- [Background] Piorkowski C, Kircher S, Arya A, Gaspar T, Esato M, Riahi S, Bollmann A, Husser D, Staab C, Sommer P, Hindricks G. Computed tomography model-based treatment of atrial fibrillation and atrial macro-re-entrant tachycardia. Europace. 2008 Aug;10(8):939-48. doi: 10.1093/europace/eun147. Epub 2008 Jun 23. PMID 18577508
- [Background] Kistler PM, Earley MJ, Harris S, Abrams D, Ellis S, Sporton SC, Schilling RJ. Validation of three-dimensional cardiac image integration: use of integrated CT image into electroanatomic mapping system to perform catheter ablation of atrial fibrillation. J Cardiovasc Electrophysiol. 2006 Apr;17(4):341-8. doi: 10.1111/j.1540-8167.2006.00371.x. PMID 16643352
- [Background] Kistler PM, Rajappan K, Jahngir M, Earley MJ, Harris S, Abrams D, Gupta D, Liew R, Ellis S, Sporton SC, Schilling RJ. The impact of CT image integration into an electroanatomic mapping system on clinical outcomes of catheter ablation of atrial fibrillation. J Cardiovasc Electrophysiol. 2006 Oct;17(10):1093-101. doi: 10.1111/j.1540-8167.2006.00594.x. PMID 16989651
- [Background] Kistler PM, Rajappan K, Harris S, Earley MJ, Richmond L, Sporton SC, Schilling RJ. The impact of image integration on catheter ablation of atrial fibrillation using electroanatomic mapping: a prospective randomized study. Eur Heart J. 2008 Dec;29(24):3029-36. doi: 10.1093/eurheartj/ehn453. Epub 2008 Oct 17. PMID 18931059
- [Background] Marai I, Suleiman M, Blich M, Lessick J, Abadi S, Boulos M. Impact of computed tomography image and contact force technology on catheter ablation for atrial fibrillation. World J Cardiol. 2016 Apr 26;8(4):317-22. doi: 10.4330/wjc.v8.i4.317. PMID 27152144
- [Background] Im SI, Shin SY, Na JO, Kim YH, Choi CU, Kim SH, Kim JW, Kim EJ, Han SW, Rha SW, Park CG, Seo HS, Oh DJ, Hwang C, Lim HE. Usefulness of neutrophil/lymphocyte ratio in predicting early recurrence after radiofrequency catheter ablation in patients with atrial fibrillation. Int J Cardiol. 2013 Oct 9;168(4):4398-400. doi: 10.1016/j.ijcard.2013.05.042. Epub 2013 May 28. No abstract available. PMID 23725815
- [Background] Ha AC, Wijeysundera HC, Birnie DH, Verma A. Real-world outcomes, complications, and cost of catheter-based ablation for atrial fibrillation: an update. Curr Opin Cardiol. 2017 Jan;32(1):47-52. doi: 10.1097/HCO.0000000000000348. PMID 27755137